CLINICAL TRIAL: NCT01260454
Title: The Qutenza® Patch for Disabling Treprostinil Infusion Site Pain
Brief Title: The Qutenza Patch as Treatment for Disabling Treprostinil (Remodulin) Infusion Site Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: United Therapeutics (Industry)
Responsible Party: Principal Investigator, R. James White, Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Qutenza White
Record Dates: First submitted 2010-12-09; First posted 2010-12-15 (Estimated); Results first posted 2016-02-22 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-03

CONDITIONS: Pulmonary Hypertension; Pulmonary Arterial Hypertension
Keywords: Qutenza; Capsaicin; Remodulin; Treprostinil
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension | interventions — Capsaicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Qutenza patch (Experimental): All participants actively treated with Qutenza
  Interventions: Drug: Qutenza (8% capsaicin)

INTERVENTIONS:
Drug: Qutenza (8% capsaicin) — We will place a Qutenza (8% capsaicin) patch onto an area of normal, anesthetized skin for 60 minutes. Within 28 days, subjects will place a new treprostinil infusion site into the area of Qutenza pre-treated skin.
  Other Names: Qutenza; Capsaicin

SUMMARY:
Subcutaneous treprostinil (Remodulin) is effective therapy for pulmonary arterial hypertension, a life threatening disease of the lung blood vessels. Unfortunately, treprostinil is irritating to the skin and many patients experience intense pain at the infusion site for the first 7-10 days after placing a new subcutaneous infusion site.

Qutenza is an FDA approved formulation of 8% capsaicin that is approved for the treatment of post-herpetic neuralgia, a painful skin condition. The investigators hypothesize that pretreatment of an area of skin with Qutenza would decrease the pain associated with a new treprostinil infusion site. The investigators hope that Qutenza will decrease both the intensity of the pain and the duration of the pain after patients place a new treprostinil infusion site.

In this initial study, the investigators will provide Qutenza in open-label, unblinded fashion and ask patients to rate their pain using a diary tool with which they are already comfortable.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary Hypertension
* Using subcutaneous treprostinil
* Already participating as a subject in our prospective study of infusion site pain
* Has documented debilitating pain (6/10 or greater) in the study after a site change

Exclusion Criteria:

* Uncontrolled hypertension
* Recent stroke or myocardial infarction

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-11; Primary Completion 2011-12 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R James White, MD, PhD, Principal Investigator — University of Rochester
Locations (1):
- Mary M. Parkes Asthma Center, University of Rochester, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 26 participants who were previously recruited for a study called "SubQ works" were screened for this study.
Pre-assignment Details: Of the 26 screened 10 had a pain score > or = 6 on two consecutive days. 6 of these 10 agreed to enroll.
Groups:
- Qutenza Patch: We will place a Qutenza patch following the package insert (60 minute application following topical anesthetic) onto an area of healthy skin. Within 28 days, subjects will place a new treprostinil infusion site into the area of Qutenza pre-treated skin.
  Qutenza (8% capsaicin): We will place a Qutenza (8% capsaicin) patch onto an area of normal, anesthetized skin for 60 minutes
Period: Overall Study
Arm/Group | Qutenza Patch
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Qutenza Patch
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 6
mean pain level [Mean (Standard Deviation); unit: Visual Analogue Scale] — Average pain over the 14 day diary period; measured by visual analog score. Pain was measured on a 10 point visual analog score with the word 'none' at 0 and 'agonizing' at 10.
  Visual Analogue Scale | 4.15 (0.85)
mean worst pain level [Mean (Standard Deviation); unit: Visual Analogue Scale] — Worst pain was defined as the highest pain experienced on any day over the 14 day diary period; measured by visual analog score. Pain was measured on a 10 point visual analog score with the word 'none' at 0 and 'agonizing' at 10.
  Visual Analogue Scale | 7.99 (1.83)
Pain Relief Experienced with as needed Analgesics [Mean (Standard Deviation); unit: units on a scale] — average pain relief perceived after using prescribed analgesics over the 14 day diary period; measured by non-continuous, qualitative word scale (0= no relief, 1= a little, 2=some, 3=a lot and 4= complete relief)
  units on a scale | 1.66 (0.86)

OUTCOME MEASURES:

1. Primary Outcome: Pain Score on a Visual Analogue Scale
Description: Patients will record the maximum intensity of pain (0-10) each day after placing an infusion site in a diary with which they are already comfortable. They will record the score each day for 14 days unless they have recorded "0" for two consecutive days.
  The primary outcome measure will be the average of those 14 maximum intensity pain scores (the sum of the maximum for each day divided by the number of days, generally 14; range 0-10).
Time Frame: 14 days after a new infusion site
Population: One subject did not meet the inclusion criteria and was excluded from the efficacy analysis.
Measure: Mean (Standard Deviation); unit: Visual Analogue Scale
Arm/Group | Qutenza Patch
Number analyzed (Participants) | 5
Visual Analogue Scale | 2.89 (0.71)
Statistical Analysis 1: Comparison: Qutenza Patch; This is open-label, uncontrolled data; the comparison is made between each individual's baseline; Test type: Superiority or Other; p = 0.03, t-test, 2 sided

2. Secondary Outcome: Number of Participants Who Experienced Greater Than 6 Pain Level Using the 10 Point Visual Analog Score
Description: Qutenza has not previously been used in patients with normal, healthy skin. We will assess the reaction to capsaicin in these patients as compared to the patients with unhealthy skin (post-herpetic neuralgia) who were studied in the registration trials for Qutenza. Pain immediately following Qutenza application was measured on a 10 point visual analog score with the word 'none' above 0 and 'agonizing' above 10.
Time Frame: 60 minute period of patch application and subsequent 3 days
Measure: Number; unit: participants
Arm/Group | Qutenza Patch
Number analyzed (Participants) | 6
participants | 3

3. Secondary Outcome: Number of Participants Who Used of Narcotics Following a Treprostinil Infusion Site Change
Description: We counted the number of participants who used any amount of narcotic during the 14 day diary period.
Time Frame: 14 days
Population: One subject did not meet the inclusion criteria and was excluded from the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Qutenza Patch
Number analyzed (Participants) | 5
participants | 4

ADVERSE EVENTS:
Arm/Group | Qutenza Patch
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 4/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Qutenza Patch (N=6)
pain at the application site (General disorders) | 3
headache (Nervous system disorders) | 1
nasal congestion (Infections and infestations) | 1
sore throat (Infections and infestations) | 1
hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes